CLINICAL TRIAL: NCT00746343
Title: Reducing Medical Risks in Individuals With Bipolar Disorder - Full Study
Acronym: MedRisk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO08020071; R01MH081003 (NIH)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I Disorder; Medical Risks; Integrated Risk Reduction Intervention; Currently in Remission; BMI

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IRRI (Experimental): The integrated risk reduction intervention (IRRI) consists of three components:
  1. psychiatric treatment by a study psychiatrist
  2. assessment, referral, monitoring, and coordination by a certified registered nurse practitioner (CRNP) of medical treatment provided by the subject's own primary care physician
  3. a healthy lifestyle behaviors program delivered by a lifestyle coach. The treating psychiatrist will work in collaboration with a CRNP and a lifestyle coach. The CRNP will assess and monitor the subject's medical needs and refer the subject to their primary care physician for care and will follow-up on adherence to the medical treatment recommendations. The CRNP will be responsible for coordinating the psychopharmacological care provided by the psychiatrist, the healthy lifestyle behaviors program that will be delivered by the lifestyle coach, and the medical care provided by the subject's PCP.
  Interventions: Behavioral: IRRI
- PCCM (Experimental): Psychiatric Care with Medical Monitoring (PCMM)
  The psychiatric care with medical monitoring condition (PCMM) consists of two components:
  1. psychiatric treatment by a study psychiatrist
  2. assessment and referral by a psychiatric research nurse for medical treatment provided by the subject's own primary care physician.
  The treating psychiatrist will be assisted by a psychiatric nurse clinician who will assess and monitor the subject's medical needs and refer the subject to their primary care physician for care.
  Interventions: Behavioral: PCCM

INTERVENTIONS:
Behavioral: IRRI — Subjects will remain in their assigned treatment condition for 24 months. IRRI subjects will meet with the lifestyle coach 25-27 times throughout the duration of the study.
  Other Names: Integrated Risk Reduction Intervention
  Arms: IRRI
Behavioral: PCCM — Subjects will remain in their assigned treatment condition for 24 months.
  Other Names: Psychiatric care with medical monitoring condition
  Arms: PCCM

SUMMARY:
The primary aim of this project is to understand whether it is possible to reduce medical risk factors in adults with bipolar disorder and, in doing so, to improve psychiatric and functional outcomes. We will examine the role of behavioral risk factors and presumed behavioral mediators and moderators of health risk in individuals suffering from bipolar I disorder. The investigators will employ an innovative behavioral intervention with guideline based psychiatric care ( Integrated Risk Reduction Intervention - IRRI) in order to target modifiable medical risk factors.

DETAILED DESCRIPTION:
IRRI is aimed at improving sleep/wake and social rhythm disturbance and achieving modest weight reduction by increasing physical activity and improving nutrition and dietary habits, while at the same time providing optimal psychiatric care and medical monitoring. This will allow us to investigate the role that improvements in sleep/wake and social rhythm regularity, diet, and physical activity have in improving psychiatric and functional outcomes. In order to examine another set or possible pathways (i.e., that it is the amelioration or psychiatric symptoms that leads to the improvements in physical health), we will contrast outcomes of subjects receiving IRRI with those of subjects receiving psychiatric care with medical monitoring (PCMM), which incorporates the same optimal psychiatric care plus monitoring of medical conditions. These aims will be achieved in a 24-month randomized treatment trial of 144 adult subjects with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 55 years
2. Body mass index (BMI) >25
3. Meets DSM-IV criteria for lifetime bipolar I disorder
4. Is in remission (with possible sub-threshold symptoms), i.e., as a HRDS-25 < or equal to 10, YMRS < or equal to 8, and CGI-BP-S <3 for two weeks
5. Able to give basic informed consent
6. Current diagnosis or past history of anxiety disorder, eating disorder, or other psychiatric comorbidities will not be exclusion criteria for participation, except those listed in the exclusion criteria below

Exclusion Criteria:

1. Ultra-rapid cycling (>8 episodes per year) bipolar I disorder
2. Presence of pervasive developmental disorder, antisocial personality disorder, current substance dependence or abuse, and organic mental disorder
3. Unstable and severe medical illness that requires immediate and intensive medical attention, for instance, a subject with a terminal illness or a subject with severe and unstabilized coronary artery disease; these subjects will be immediately referred to the most appropriate medical and psychiatric treatment. When appropriate, the subjects can be reconsidered for inclusion in the study if/when their medical condition becomes compatible with participation in a protocol-driven research study
4. Unwilling or unable to comply with study requirements (i.e., complete forms, attend scheduled evaluations)
5. Not competent to provide informed consent in the opinion of the investigator
6. Women who are planning to become pregnant, currently pregnant, or breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2008-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Integrated risk reduction intervention (IRRI), compared with psychiatric care with medical monitoring, will result in a larger decrease in medical risk factors and a greater improvement in sleep/wake and social rhythm disturbances. | Entry and every 6 months of participation for two years
Integrated risk reduction intervention compared with psychiatric care with medical monitoring will result in greater improvement in mood symptoms and functioning, particularly employment-related functioning. | Entry and every 6 months of participation for two years

SECONDARY OUTCOMES:
The effect of integrated risk reduction intervention on improved mood symptoms and functioning will be mediated by the effect of integrated risk reduction intervention on medical risk factors and on sleep/wake and social rhythm disturbances. | 6, 12, and 18 month timepoints of participation
In turn, the effect of integrated risk reduction intervention on medical risk factors and on sleep/wake and social rhythm disturbances will be mediated by the regular participation and adherence of the subject to integrated risk reduction intervention. | This is assessed by how many missed appointments the subject has for IRRI

CONTACTS AND LOCATIONS:
Overall Officials: David J Kupfer, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States